CLINICAL TRIAL: NCT01932268
Title: A Pilot Study for Pharmacokinetic Parameter of Colchicine in Patient Taking Rifampin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Colchicine_RFP 2011_1
Record Dates: First submitted 2011-12-07; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Kidney Disease; Tuberculosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Tuberculosis | interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rifampicin (Experimental): experimentally check a change of the colchicine concentration from baseline at 1,2,4,8,24 hours after taking Rifampicin
  Interventions: Drug: Rifampicin

INTERVENTIONS:
Drug: Rifampicin — single arm : check a change of Colchicine concentrations from basline at 1,2,4,8,24 hours after Rifampicin administration
  Other Names: Rifampin

SUMMARY:
The purpose of this study is to examine the colchicine concentration before and after the administration of rifampicin.

ELIGIBILITY:
Inclusion Criteria:

* from 18yrs to 80yrs , man and women
* the patient who are taking rifampicine over 2weeks
* the patient sign on the concent form

Exclusion Criteria:

* the patient have experience to take medication that have an effect on renal function
* the patient have hypersensitivity to colchicine
* At least, the average level of two separate blood pressure ( 2min interval ) shows that SBP <= 100 mmHg or >=160 mmHg and DBP <=60 mmHg >=100 mmHg, or Heart rate < 40 beats/min or > 90 beats/min
* uncontrolled hypertension
* serum albumin < 3.5, > 5 g/dL
* acute hepatitis or the level of AST or ALT is over 2times of normal range or the level of bilirubin is over 2.0 mg/dL
* the patient who have gastro-intestinal disease ( ex, crohn's disease, acute or chronic pancreatitis, ulcer )or who have the surgical history of gastrointestine.
* the patient who should take azathioprine, mercaptopurine, cyclophosphamide, Losartan, benzbromarone,fenofibrate,furosemide ,probenecid
* the patient who had taken part in the other study within 3months
* the patient who had gotten blood transfusion
* pregnant, breast feeding

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
a change of the colchicine concentration from baseline at 1,2,4,8,24 hours after Rifampicin administration | the colchicine concentration of baseline(C0) and at 1(C1),2(C2),4(C4),8(C8),24(C24) hours after Rifampicin administration